CLINICAL TRIAL: NCT05687084
Title: Randomized Controlled Trial on the Oncologic Outcomes of Use Versus Not Use of the Uterine Manipulator in the Surgical Treatment of Apparent Uterine-confined Endometrial Carcinoma
Brief Title: Uterine Manipulator Versus No Uterine Manipulator in Endometrial Cancer Trial
Acronym: MANEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Stefano Uccella, Prof. Stefano Uccella, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MANEC Trial
Record Dates: First submitted 2022-11-06; First posted 2023-01-17 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Neoplasms
Keywords: Endometrial Neoplasms; Uterine manipulator; Laparoscopic hysterectomy; Recurrence-free survival; Cause-specific survival; Overall survival; Oncologic outcomes
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicenter, parallel arms, open-label, randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total hysterectomy with a uterine manipulator (Experimental): Total hysterectomy with bilateral salpingo-oophorectomy performed with the use of a uterine manipulator during surgery.
  Interventions: Device: Uterine manipulator use
- Total hysterectomy without a uterine manipulator (No Intervention): Total hysterectomy with bilateral salpingo-oophorectomy performed without the use of a uterine manipulator during surgery.

INTERVENTIONS:
Device: Uterine manipulator use — The uterine manipulator will be inserted into the uterus to assist in the procedure of total hysterectomy.
  Arms: Total hysterectomy with a uterine manipulator

SUMMARY:
Minimally invasive surgery is the recommended approach in endometrial cancer (EC) patients based on the results of two randomized controlled trials, given its advantages without compromised oncologic outcomes. The uterine manipulator is commonly used in benign and malignant pathologies to perform a laparoscopic or robotic hysterectomy. However, although regularly used, the uterine manipulator adoption in EC is a controversial technical aspect due to the raised concerns regarding the possible risk of disruption of the tumor mass, the spread of malignant cells, and seeding of the disease, particularly at the level of the vaginal cuff or spread of tumor cells, with increased risk of recurrence and death due to EC. On that basis, given that hysterectomy without a uterine manipulator is feasible, only a randomized controlled trial comparing oncologic outcomes in EC patients after use versus not use of the uterine manipulator will be able to provide high-quality evidence to answer this critical question and allow or exclude the use of a uterine manipulator during minimally invasive hysterectomy for EC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Endometrial Cancer of any histology (including carcinosarcoma) and grade
* Planned surgical treatment including hysterectomy and bilateral salpingo-oophorectomy (ovarian preservation in selected patients is not an exclusion criterion)
* Age ≥ 18 years
* No preoperative evidence of extrauterine disease (Clinical stage IIIA, IIIB)
* No preoperative evidence of suspicious lymph nodes (Clinical stage IIIC)
* No preoperative evidence of distant metastasis (Clinical stage IV)
* Approved and signed informed consent

Exclusion Criteria:

* Neoadjuvant therapy
* Synchronous or previous (< 5 years) invasive cancer, not including non-melanoma skin cancer
* Fertility preservation
* World Health Organization performance score > 2
* Uterine sarcoma
* Previous pelvic/abdominal radiotherapy, hormone therapy for cancer (< 5 years), chemotherapy (< 5 years), pelvic or paraaortic lymphadenectomy, or retroperitoneal surgery
* Inadequate bone marrow function (white blood cells <3·0×109/L, platelets <100×109/L)
* Inadequate liver function (bilirubin >1.5×upper normal limit [UNL], aspartate aminotransferase, and alanine aminotransferase >2.5 × UNL)
* Inadequate kidney function (creatinine clearance < 60 mL per min calculated according to Cockcroft-Gault 10 or < 50 mL per min Ethylenediaminetetraacetic acid clearance)
* Intraoperative evidence of stage IV disease

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | Each follow-up visit, up to 4 years from the day of surgery
  Any recurrence or death related to endometrial cancer (EC) or treatment

SECONDARY OUTCOMES:
Cause-specific survival | Each follow-up visit, up to 4 years from the day of surgery
  Any death related to endometrial cancer (EC) or treatment
Overall survival | Each follow-up visit, up to 4 years from the day of surgery
  Any death for any cause
Site-specific recurrence-free survival | Each follow-up visit, up to 4 years from the day of surgery
  Any recurrence per site of first recurrence
Operative time | Day of surgery
  Time between first incision and skin closure
Intraoperative blood loss | Day of surgery
  Total blood aspirate during the surgical procedure
30-day post-surgical morbidity | 30 days after surgery
  Perioperative (intraoperative and postoperative) complications graded based on the Clavien-Dindo classification
Lymphovascular space invasion | Day of surgery
  Presence of lymphovascular space invasion at definitive pathology
Peritoneal cytology | Day of surgery
  Presence of positive peritoneal cytology at definitive pathology
Quality of life indexes | Each follow-up visit, up to 4 years from the day of surgery
  The Functional Assessment of Cancer Therapy - General (FACT-G) - A 27-item questionnaire designed to measure four domains of Health-Related Quality of Life in cancer patients: Physical, social, emotional, and functional well-being. Score range 0-108. The higher the score, the better the Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Uccella, MD, PhD, Principal Investigator — AOUI Verona - University of Verona; Simone Garzon, MD, Principal Investigator — AOUI Verona - University of Verona; Pier Carlo Zorzato, MD, Principal Investigator — AOUI Verona - University of Verona
Locations (3):
- Italy (3):
  - UOC Ostetricia e Ginecologia, Azienda Ospedaliera Santa Croce e Carle, Cuneo, Italy
  - UOC Ostetricia e Ginecologia, Arcispedale Santa Maria Nuova, Reggio Emilia
  - AOUI Verona - University of Verona - Department of Obstetrics and Gynecology, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Concin N, Matias-Guiu X, Vergote I, Cibula D, Mirza MR, Marnitz S, Ledermann J, Bosse T, Chargari C, Fagotti A, Fotopoulou C, Gonzalez Martin A, Lax S, Lorusso D, Marth C, Morice P, Nout RA, O'Donnell D, Querleu D, Raspollini MR, Sehouli J, Sturdza A, Taylor A, Westermann A, Wimberger P, Colombo N, Planchamp F, Creutzberg CL. ESGO/ESTRO/ESP guidelines for the management of patients with endometrial carcinoma. Int J Gynecol Cancer. 2021 Jan;31(1):12-39. doi: 10.1136/ijgc-2020-002230. Epub 2020 Dec 18. PMID 33397713
- [Background] van den Haak L, Alleblas C, Nieboer TE, Rhemrev JP, Jansen FW. Efficacy and safety of uterine manipulators in laparoscopic surgery: a review. Arch Gynecol Obstet. 2015 Nov;292(5):1003-11. doi: 10.1007/s00404-015-3727-9. Epub 2015 May 13. PMID 25967852
- [Background] Uccella S, Cianci S, Gueli Alletti S. Uterine manipulator in endometrial cancer: we are still far from the answer. Am J Obstet Gynecol. 2021 Mar;224(3):332. doi: 10.1016/j.ajog.2020.09.049. Epub 2020 Nov 15. No abstract available. PMID 33207238
- [Background] Uccella S, Bonzini M, Malzoni M, Fanfani F, Palomba S, Aletti G, Corrado G, Ceccaroni M, Seracchioli R, Shakir F, Ferrero A, Berretta R, Tinelli R, Vizza E, Roviglione G, Casarella L, Volpi E, Cicinelli E, Scambia G, Ghezzi F. The effect of a uterine manipulator on the recurrence and mortality of endometrial cancer: a multi-centric study by the Italian Society of Gynecological Endoscopy. Am J Obstet Gynecol. 2017 Jun;216(6):592.e1-592.e11. doi: 10.1016/j.ajog.2017.01.027. Epub 2017 Jan 29. PMID 28147240
- [Background] Padilla-Iserte P, Lago V, Tauste C, Diaz-Feijoo B, Gil-Moreno A, Oliver R, Coronado P, Martin-Salamanca MB, Pantoja-Garrido M, Marcos-Sanmartin J, Gilabert-Estelles J, Lorenzo C, Cazorla E, Roldan-Rivas F, Rodriguez-Hernandez JR, Sanchez L, Muruzabal JC, Hervas D, Domingo S; Spanish Society of Gynecology and Obstetrics Spanish Investigational Network Gynecologic Oncology Group. Impact of uterine manipulator on oncological outcome in endometrial cancer surgery. Am J Obstet Gynecol. 2021 Jan;224(1):65.e1-65.e11. doi: 10.1016/j.ajog.2020.07.025. Epub 2020 Jul 18. PMID 32693096
- [Derived] Uccella S, Puppo A, Ghezzi F, Zorzato PC, Ceccaroni M, Mandato VD, Berretta R, Camanni M, Seracchioli R, Perrone AM, Chiantera V, Vizzielli G, Sozzi G, Beretta P, Steinkasserer M, Legge F, Stevenazzi G, Candotti G, Bergamini V, Fanfani F, Garzon S. A randomized controlled trial on the oncologic outcomes of use of the intrauterine manipulator in the treatment of apparent uterine-confined endometrial carcinoma: the MANEC Trial. Int J Gynecol Cancer. 2024 Dec 2;34(12):1971-1975. doi: 10.1136/ijgc-2024-005668. PMID 39266205